CLINICAL TRIAL: NCT04096040
Title: Benefits of Microcor in Ambulatory Decompensated Heart Failure
Acronym: BMAD-TX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 90D0202
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device Data Engagement Assessment (Experimental): This arm will assess the endpoints of investigator engagement with the device data.
  Interventions: Device: μCor

INTERVENTIONS:
Device: μCor — μCor consists of the following components: A) Patch B) Sensor C) Charger D) Data transmission device (Gateway) E) Server Once activated, the wearable Sensor automatically acquires ECG, RF readings, heart rate, respiration rate, activity, and posture measurements.

SUMMARY:
To assess investigator engagement of μCor system data in the context of heart failure management. The μCor system includes a sensor and wearable patch for fluid management.

DETAILED DESCRIPTION:
Subjects meeting the inclusion/exclusion criteria will wear the μCor for up to 90 days.

During the study, face to face follow up will occur every 30 days. For all subjects, each scheduled clinic visit will include assessment of cardiac signs, symptoms, and any relevant clinically actionable events.

The subject will be given a daily diary to track symptoms, hospital visits, medication changes, and all other heart failure related clinical events.

Weekly phone calls to the subject will be given throughout the duration of the study to remind the patient to use the subject diary and to collect and record heart failure related clinical events.

The subject's health care provider team will receive the μCor data through access to a clinical tool interface. The clinical tool will send data updates that are dependent on the μCor data trends. The data updates will allow the health care provider team to take action when the data indicate worsening heart failure, within the context of standard of care medical practice and patient specific parameters. Weekly data reports will be delivered to the investigators.

Subjects will be contacted six months and one year from initial enrollment to assess the vital status of the subject, any heart failure related clinical events since the end of μCor wear, and any health care utilization since the end of μCor wear.

ELIGIBILITY:
Inclusion Criteria:

* 4.1.1 Subjects hospitalized for acute decompensated heart failure and enrolled in the study within 10 days post-hospital discharge.
* 4.1.2 Subjects who have had an acute heart failure event requiring medical management in the previous 180 days of index hospitalization admission. This acute heart failure event admission must be at least 2 weeks apart from the event admission in 4.1.1
* 4.1.3 Subjects 21 years of age or older on the day of screening.

Exclusion Criteria:

* 4.2.1 Subjects who are wearing the wearable cardioverter defibrillator (WCD)
* 4.2.2 Subjects not expected to survive one year from enrollment from non-cardiac disease.
* 4.2.3 Subjects with skin allergy or sensitivity to medical adhesives.
* 4.2.4 Subjects anticipated to start dialysis within 90 days.
* 4.2.5 Subjects currently implanted with an subcutaneous implantable cardio defibrillator (S-ICD) system.
* 4.2.6 Subjects who received a percutaneous coronary intervention (PCI) less than 24 hours after onset of heart failure related symptoms during index hospitalization.
* 4.2.7 Subjects who are unable to participate in all follow up visits.
* 4.2.8 Subjects participating in research other than a registry at the time of enrollment.
* 4.2.9 Subjects currently implanted with a Left Ventricular Assist Device (LVAD).
* 4.2.10 Subjects with self-reported pregnancy.
* 4.2.11 Subjects currently being actively managed with any device based remote HF monitoring.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Osz, Study Director — Zoll Medical Corporation
Locations (80):
- United States (67):
  - SYED Research Consultants LLC, Sheffield, Alabama
  - TriWest Research, El Cajon, California
  - Zillan Clinical Research, Inglewood, California
  - Axis Clinical Trials, Los Angeles, California
  - InvivoCure LLC, Mission Hills, California
  - ACRC Studies, San Diego, California
  - Aventura Clinical Research LLC, Aventura, Florida
  - Accel Research Sites - Guardian, Davenport, Florida
  - Accel Research Sites- Daytona Heart Group, DeLand, Florida
  - Accel Research Sites - Guardian Winter Park, Deltona, Florida
  - Holy Cross Hospital, Medical Group, Cardiology Associates, Fort Lauderdale, Florida
  - Elite Cardiac Research Center, Hialeah, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Homestead Associates in Research, Miami, Florida
  - Westchester Research Center at Westchester General Hospital, Miami, Florida
  - Miramax Clinical Research Inc, North Miami, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Accel Research Sites, Orlando, Florida
  - DBC Research, Tamarac, Florida
  - Winter Haven Hospital - BayCare Health System, Winter Haven, Florida
  - Accel Research Sites - Guardian Winter Park, Winter Park, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Columbus Cardiology Associates, Columbus, Georgia
  - Accel Research Sites - Lake County Medical Group, Eatonton, Georgia
  - Quincy Medical Group, Quincy, Illinois
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Beacon Medical Group, South Bend, Indiana
  - Norton Heart Specialists, Louisville, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Sinai Center for Thrombosis Reserach and Drug Development, Baltimore, Maryland
  - Intervent Clinical Research Center, Pembroke Hills, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Ascension Providence Rochester Hospital, Rochester, Michigan
  - Ascension St. Mary's Research Institute, Saginaw, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Kansas City Cardiology, Lee's Summit, Missouri
  - Gateway Cardiovascular Research Center, Inc, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Methodist Physicians Clinical Heart Consultants, Omaha, Nebraska
  - Virtua Health, Cherry Hill, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Bassett Medical Center, Cooperstown, New York
  - Laurelton Heart Specialist, Rosedale, New York
  - BronxCare Health System at BronxCare Hospital Center, The Bronx, New York
  - Macklenberg Heart Specialists / Focus Clinical Research Solutions, Charlotte, North Carolina
  - Heart House Research Foundation, Springfield, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Mercer Bucks Cardiology at Jefferson Health, Newtown, Pennsylvania
  - Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Knoxville HMA Cardiology, PPM, LLC, Knoxville, Tennessee
  - North Texas Research Associates, Allen, Texas
  - North Houston Cardiology Center, Cypress, Texas
  - JPS Health Network, Fort Worth, Texas
  - North Texas Research Associates, McKinney, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Mission Research Institue, New Braunfels, Texas
  - Bay Area Heart, Webster, Texas
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Pulse Heart Institute, Puyallup, Washington
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Klinik Favoriten, Vienna
- France (4):
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Cardiologique, Lille
  - CHU Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Chu Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Hôpital Européen Georges Pompidou - Centre d'Investigations Cliniques - Pôle D - étage 5, Paris
- Germany (7):
  - Albertinen Krankenhaus HH, Hamburg, GG
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Albertinen Krankenhaus Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Herzzentrum Leipzig, Universitätsklinik für Kardiologie Abteilung Rhythmologie, Leipzig

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- uCor Wearers: Subjects wearing the uCor device
Period: Overall Study
Arm/Group | uCor Wearers
Started | 265
Completed | 249
Not Completed | 16
Not completed — Protocol Violation | 12
Not completed — Non-compliant site | 4

BASELINE CHARACTERISTICS:
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 144
Race/Ethnicity, Customized [Number; unit: participants] — Participant could identify as more than one ethnicity and may be counted in more than one ethnic category.
  participants
    American Indian or Alaskan Native | 1
    Asian | 3
    Caucasian | 135
    Black or African American | 63
    Other | 5
    Don't Know/ No Response | 0
    Hispanic/ Latino | 43
Weight [Mean (Standard Deviation); unit: pounds] | 205.2 (63.4)
Height [Mean (Standard Deviation); unit: inches] | 66.6 (4.1)
Blood Pressure (Systolic) [Mean (Standard Deviation); unit: mmHg] | 126.2 (20)
Blood Pressure (Diastolic) [Mean (Standard Deviation); unit: mmHg] | 72.2 (12.1)
Heart Rate (per min) [Mean (Standard Deviation); unit: beats per minute] | 77.1 (13.2)
Respiratory Rate (per min) [Mean (Standard Deviation); unit: breaths per minute] | 18 (5.7)
Time Since Heart Failure Diagnosis [Mean (Standard Deviation); unit: years] | 4.7 (5.8)
Ejection Fraction (Min) [Mean (Standard Deviation); unit: percent of ejection fraction] | 41.3 (15.6)
Ejection Fraction (Max) [Mean (Standard Deviation); unit: percent of ejection fraction] | 44.9 (15.7)
New York Heart Association(NYHA) Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification places patients in 1 of 4 categories based on limitations of physical activity. The healthcare practitioner assigns the patient. I= No limitation of physical activity. II= Slight limitation of physical activity. III= Marked limitation of physical activity. IV= Symptoms of heart failure at rest- Any physical activity causes further discomfort.
  Participants
    Class I | 7
    Class II | 102
    Class III | 84
    Class IV | 2
    Not Documented | 54
Heart Failure Etiology [Count of Participants; unit: Participants]
  Ischemic | 102
  Non-ischemic | 130
  Mixed | 13
  N/A or Unknown | 4
Educational Level [Count of Participants; unit: Participants]
  Less than High School | 57
  High School | 132
  Bachelors or Associates | 37
  Graduate or Professional | 13
  N/A or Unknown | 10
Employment Status [Count of Participants; unit: Participants]
  Employed | 32
  Student | 0
  Homemaker | 2
  Unemployed | 63
  Retired | 152
Cardiac Device History [Count of Participants; unit: Participants]
  History of Implantable Cardioverter Defibrillator(ICD): Yes | 49
  History of Implantable Cardioverter Defibrillator(ICD): No | 200
  History of Implantable Cardioverter Defibrillator(ICD): N/A or Unknown | 0
  ICD Active at Enrollment: Yes | 49
  ICD Active at Enrollment: No | 0
  ICD Active at Enrollment: N/A or Unknown | 200
  History of Pacemaker: Yes | 45
  History of Pacemaker: No | 204
  History of Pacemaker: N/A or Unknown | 0
  Pacemaker Active at Enrollment: Yes | 43
  Pacemaker Active at Enrollment: No | 2
  Pacemaker Active at Enrollment: N/A or Unknown | 204
History of Remote Heart Failure(HF) Monitor [Number; unit: participants]
  Yes | 2
  No | 247
History of Hypertension [Count of Participants; unit: Participants]
  Yes | 233
  No | 14
  Uknown | 2
History of Diabetes [Count of Participants; unit: Participants]
  Yes | 141
  No | 107
  Unknown | 1
History of Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  Yes | 86
  No | 157
  Unknown | 6
History of Transient Ischemic Attack (TIA) [Count of Participants; unit: Participants]
  Yes | 33
  No | 215
  Unknown | 1
History of Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants]
  Yes | 118
  No | 128
  Unknown | 3
History of Angina [Count of Participants; unit: Participants]
  Yes | 78
  No | 159
  Unknown | 12
History of Syncope [Count of Participants; unit: Participants]
  Yes | 33
  No | 208
  Unknown | 8
History of Sudden Cardiac Arrest (SCA) [Count of Participants; unit: Participants]
  Yes | 9
  No | 237
  Unknown | 3
History of Arrhythmia [Count of Participants; unit: Participants]
  Yes | 153
  No | 88
  Unknown | 8
History of Myocardial Infarction (MI) [Count of Participants; unit: Participants]
  Yes | 83
  No | 157
  Unknown | 9
History of Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants]
  Yes | 48
  No | 199
  Unknown | 2
History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants]
  Yes | 85
  No | 161
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Data Updates Received by the uCor Subject Management System
Description: Each time a subject's thoracic fluid index (TFI) exceeded a threshold for 3 consecutive days, a data update report was generated by the uCor management system. The site then confirmed its receipt of the data update by completing a case report form. At least 1 of these case report forms was completed for 56 subjects.
Time Frame: 90 days
Population: data updates per subject
Measure: Median (Inter-Quartile Range); unit: data updates per subject
Units Other Than Participants: data updates
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Number analyzed (data updates) | 415
data updates per subject | 3 [1 to 10]

2. Primary Outcome: Approximate Time Spent Reviewing Data Reports Assessment Across Sites (PO 2: Part 1/2)
Description: Sites reviewed data reports in each of the following contexts: planned weekly phone call, planned office visit, unplanned phone call, unplanned office visit, and data update. Sites reported whether they spent less than 5, 5 to 10, or greater than 10 minutes reviewing each report. At least 1 of these case report forms was completed for 214 subjects.
Time Frame: 90 days
Measure: Count of Units; unit: Number of data reports
Units Other Than Participants: Number of data reports
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Number analyzed (Number of data reports) | 2107
Number of data reports
  0-5 minutes | 1548
  5-10 minutes | 427
  >10 minutes | 132

3. Primary Outcome: Approximate Time Spent Reviewing Data Reports Assessment Within Sites (PO 2: Part 2/2)
Description: as for outcome 2
Time Frame: 90 days
Population: Most common amount of time spent reviewing by each site
Measure: Number; unit: number of sites
Units Other Than Participants: number of sites
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Number analyzed (number of sites) | 44
number of sites
  0-5 minutes | 34
  5-10 minutes | 9
  >10 minutes | 1

4. Primary Outcome: The Number of Medication Changes(MC) and Lifestyle Modifications(LS) Recommended to the Subject Based on Evaluating μCor Data and Symptoms (PO 3: Part 1/3)
Description: Sites reviewed data reports in each of the following contexts: planned weekly phone call, planned office visit, unplanned phone call, unplanned office visit, and data update. In each context, the subject was asked whether their symptoms changed. If yes, the site reported in a case report form whether it took action to treat the subject in the form of a medication change or lifestyle modification. At least one of these case report forms (CRFs) was completed for 214 subjects
Time Frame: 90 days
Population: Number of medication changes or lifestyle modifications per subject based on μCor data and symptoms
Measure: Count of Units; unit: number of MC/LS changes
Units Other Than Participants: number of MC/LS changes
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Number analyzed (number of MC/LS changes) | 159
number of MC/LS changes
  Number of medication changes based on μCor data and symptoms | 114
  Number of lifestyle modifications based on μCor data and symptoms | 45

5. Primary Outcome: The Number of Medication Changes(MC) and Lifestyle Modifications(LS) Recommended to the Subject Based on Evaluating μCor Data and Symptoms (PO 3: Part 2/3)
Description: as for outcome 4
Time Frame: 90 days
Population: Number of subjects with medication changes based on μCor data and symptoms
Measure: Count of Participants; unit: Participants
Arm/Group | uCor Wearers
Number analyzed (Participants) | 68
Participants
  Number of subjects with 1 medication change(s) based on μCor data and symptoms | 38
  Number of subjects with 2 medication change(s) based on μCor data and symptoms | 19
  Number of subjects with 3+ medication change(s) based on μCor data and symptoms | 11

6. Primary Outcome: The Number of Medication Changes(MC) and Lifestyle Modifications(LS) Recommended to the Subject Based on Evaluating μCor Data and Symptoms (PO 3: Part 3/3)
Description: as for outcome 4
Time Frame: 90 days
Population: Number of subjects with lifestyle modifications based on μCor data and symptoms
Measure: Count of Participants; unit: Participants
Arm/Group | uCor Wearers
Number analyzed (Participants) | 17
Participants
  Number of subjects with 1 lifestyle modification(s) based on μCor data and symptoms | 8
  Number of subjects with 2 lifestyle modification(s) based on μCor data and symptoms | 2
  Number of subjects with 3 lifestyle modification(s) based on μCor data and symptoms | 3
  Number of subjects with 4+ lifestyle modification(s) based on μCor data and symptoms | 4

7. Primary Outcome: The Number of Medication Changes Based on Subject Incidental Findings
Description: During weekly planned phone calls, planned office visits, and unplanned office visits, sites asked subjects whether they underwent any changes to their heart failure and/or cardiac medications since the last phone call and reported the result in a case report form. At least 1 of these case report forms was completed for 241 subjects.
Time Frame: 90 days
Population: Subjects with Medication Changes (MC) based on incidental findings
Measure: Count of Participants; unit: Participants
Arm/Group | uCor Wearers
Number analyzed (Participants) | 139
Participants
  Number of subjects with 1 medication change(s) based on incidental findings | 58
  Number of subjects with 2 medication change(s) based on incidental findings | 35
  Number of subjects with 3 medication change(s) based on incidental findings | 20
  Number of subjects with 4 medication change(s) based on incidental findings | 10
  Number of subjects with 5 medication change(s) based on incidental findings | 8
  Number of subjects with 6+ medication change(s) based on incidental findings | 8

8. Primary Outcome: Number of Times High μCor Measurements Were Reduced Below Threshold Levels After Medication Was Titrated or Lifestyle Modifications Were Recommended
Description: 482 medication changes or lifestyle (MC/LS) modifications occurred within the first 90 days of the study. To include only medication changes preceded and followed by sufficient µCor data to determine a threshold crossing, medication changes within the first 2 weeks of the study or the final 3 weeks of device wear were discarded. This resulted in in 262 analyzable changes. Changes occurring within 1 week of another change were grouped together. This resulted in 192 change events. Time windows were defined as 0-13 days before the first change in a change event vs. 8-21 days after the last change in a change event. A high μCor measurement was defined as the receipt of a data update by the site. A low μCor measurement was defined as the absence of a data update received by the site.
Time Frame: 90 days
Population: MC/LS events preceded by a high uCor measurement within -13 to 0 days
Measure: Count of Units; unit: MC/LS change events
Units Other Than Participants: MC/LS change events
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Number analyzed (MC/LS change events) | 40
MC/LS change events
  MC/LS preceded by a high μCor meas. w/i -13 to 0 days,followed by a high uCor meas. w/i +8 to+21days | 19
  MC/LS preceded by a high μCor meas. w/i -13 to 0 days,followed by a low uCor meas. w/i +8 to+21 days | 21

9. Secondary Outcome: Strength of Association Between μCor Measurements and Clinically Related Heart Failure Events.
Description: Definitions:
  Daytime: 7:00 AM - 12:00 AM Nighttime: 12:00 AM - 7:00 AM
  For each day on which the subject wore the device, the following values were calculated:
  Daytime activity: The proportion of minutes while wearing the device that the subject spent active (unitless).
  Nighttime heart rate: The median heart rate while wearing the device during the night (beats/min) Thoracic fluid index: The median proportion of ratio of radiofrequency-measured lung fluid readings compared to the subject's baseline (unitless).
  Nighttime posture: The median pitch angle while wearing the device during the night (degrees, where 0 is the horizontal).
  Nighttime respiration: The median respiration rate while wearing the device during the night (breaths/min)
  HF event: a hospitalization, emergency room visit, observation unit visit, unplanned clinic visit, or death primarily due to heart failure.
Time Frame: 90 days
Population: The median was calculated for the 7 days prior to the 1st heart failure (HF) event; the median was calculated for the final 7 days of device wear. ROC analysis was performed. Data are presented assuming that the device reading in subjects without events is less than that of subjects with events. Unit of measure: probability that a randomly chosen subject with severe symptoms has a greater device value than a randomly chosen subject with mild symptoms.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
probability
  Nighttime Heart Rate | 0.57 [0.45 to 0.68]
  Nighttime Respiration Rate | 0.52 [0.39 to 0.66]
  Nighttime Posture | 0.57 [0.46 to 0.68]
  Thoracic Fluid Index | 0.61 [0.51 to 0.71]
  Daytime Activity | 0.45 [0.34 to 0.57]

10. Secondary Outcome: Strength of Association Between μCor Measurements and Subject Reported Symptoms
Description: During office visits at months 1, 2, and 3, subjects reported their degrees of dyspnea, orthopnea, and fatigue on the following scale: [none, seldom, frequent, continuous]. Each day that the subject wore the device, a daily median was calculated for the following measures: [thoracic fluid index, nighttime heart rate, nighttime respiration rate]. Nighttime was defined as 12:00 AM - 7:00 AM.
Time Frame: 90 days
Population: The median of the daily medians for each device measure was calculated for the 7 days preceding each office visit. To assess whether reports of severe [frequent or continuous] symptoms were associated with greater device measures than reports of mild symptoms [none or seldom], ROC analysis was performed. Unit of measure: probability that a randomly chosen subject with severe symptoms has a greater device value than a randomly chosen subject with mild symptoms.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
probability
  Dyspnea and Thoracic Fluid Index (TFI) | 0.54 [0.47 to 0.61]
  Dyspnea and Nighttime Heart Rate | 0.49 [0.42 to 0.56]
  Dyspnea and Nighttime Respiration Rate | 0.52 [0.45 to 0.59]
  Orthopnea and Thoracic Fluid Index (TFI) | 0.52 [0.44 to 0.61]
  Orthopnea and Nighttime Heart Rate | 0.53 [0.44 to 0.62]
  Orthopnea and Nighttime Respiration Rate | 0.60 [0.52 to 0.69]
  Fatigue and Thoracic Fluid Index (TFI) | 0.57 [0.50 to 0.63]
  Fatigue and Nighttime Heart Rate | 0.51 [0.45 to 0.58]
  Fatigue and Nighttime Respiration Rate | 0.54 [0.48 to 0.61]

11. Secondary Outcome: Correlations Between uCor Measurements and Patient Reported Symptoms: Mild/Severe Symptoms
Description: During office visits at months 1, 2, and 3, subjects reported their degrees of dyspnea, orthopnea, and fatigue on the following scale: [none, seldom, frequent, continuous].
Time Frame: 90 days
Population: Each of the 249 participants in the study could contribute data to either Arm/Group depending on the severity of their symptoms across the 3-month study duration.
Measure: Number; unit: Symptom reports
Groups:
- uCor Wearers Reporting Mild Symptoms: Subjects wearing the uCor device that reported mild symptoms that were preceded by a valid device measure.
- uCor Wearers Reporting Severe Symptoms: Subjects wearing the uCor device that reported severe symptoms that were preceded by a valid device measure.
Arm/Group | uCor Wearers Reporting Mild Symptoms | uCor Wearers Reporting Severe Symptoms
Number analyzed (Participants) | 249 | 249
Symptom reports
  Dyspnea - Thoracic Fluid Index (TFI) | 255 | 100
  Dyspnea - Nighttime Heart Rate (NHR) | 253 | 99
  Dyspnea - Nighttime Respiration Rate (NRR) | 254 | 99
  Orthopnea - Thoracic Fluid Index (TFI) | 299 | 56
  Orthopnea - Nighttime Heart Rate (NHR) | 294 | 57
  Orthopnea - Nighttime Respiration Rate (NRR) | 296 | 56
  Fatigue - Thoracic Fluid Index (TFI) | 232 | 123
  Fatigue - Nighttime Heart Rate (NHR) | 227 | 124
  Fatigue - Nighttime Respiration Rate (NRR) | 230 | 122

12. Secondary Outcome: Hospital Readmission Rate, Physician Visit Rate, and Outpatient Clinic Visit Rate During the Study Period
Description: For each weekly phone call and monthly office visit, each subject reported whether they experienced a hospitalization or emergency room visit since their last call/visit. An adjudication committee of physicians determined whether each event was due to HF or not.
Time Frame: 90 days
Population: Subjects who had hospital readmission, physician visit, and/or outpatient clinic visit during the study period
Measure: Count of Participants; unit: Participants
Arm/Group | uCor Wearers
Number analyzed (Participants) | 39
Participants
  Subjects with Hospital Readmission for Heart Failure between enrollment and Day 90 | 32
  Subjects with an ER visit for Heart Failure between enrollment and Day 90 | 7

13. Secondary Outcome: Mortality Rate, Heart Failure Related Events, Quality of Life (QoL) and Healthcare Utilization Data at 6 Months and One Year Post Enrollment: Mortality Data
Description: On each subject's final date of study participation, their survival status was recorded.
Time Frame: 6 months and 1 year
Population: Descriptive statistics around mortality rate, cause of death, quality of life (QoL), and health care utilization among patients six months and one year after enrollment into the study.
Measure: Count of Participants; unit: Participants
Groups:
- uCor Wearers - 6 Month Data: Subjects still active in the study at 6 months post-enrollment
- uCor Wearers - 1 Year Data: Subjects still active in the study at 1 year post-enrollment.
Arm/Group | uCor Wearers - 6 Month Data | uCor Wearers - 1 Year Data
Number analyzed (Participants) | 249 | 249
Participants
  Number of Subjects reported as deceased | 20 | 37
  Number of Subjects not reported as deceased | 229 | 212

14. Secondary Outcome: Mortality Rate, Cause of Death, Quality of Life (QoL) and Healthcare Utilization Data at 6 Months and One Year Post Enrollment: Cause of Death
Description: On each subject's final date of study participation, in the case of death, the cause of death was recorded.
Time Frame: 6 months and 1 year
Population: as for outcome 13
Measure: Number; unit: Deaths
Units Other Than Participants: Deaths
Arm/Group | uCor Wearers
Number analyzed (Participants) | 249
Number analyzed (Deaths) | 37
Deaths
  Cardiac-Sudden Cardiac Arrest | 2
  Cardiac-Heart Failure | 10
  Cardiac-Hypotension | 1
  Cardiac-Heart Disease | 1
  Non-cardiac | 12
  Unknown | 11

15. Secondary Outcome: Mortality Rate, Heart Failure Related Events, Quality of Life (QoL) and Healthcare Utilization Data at 6 Months and One Year Post Enrollment: Quality of Life Data
Description: At 0 months, 6 months, and 1 year after enrollment, subjects completed a Kansas City Cardiomyopathy Questionnaire (KCCQ-12). Quality of life is calculated as:
  KCCQ12-QL = 100*[(average of Questions 6 and 7) - 1]/4 Score is scaled 0-100, where 0 denotes the lowest reportable health status and 100 the highest.
Time Frame: 6 months and 1 year
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- uCor Wearers - Baseline: Subjects wearing the uCor device who were enrolled appropriately into the study
Arm/Group | uCor Wearers - Baseline | uCor Wearers - 6 Month Data | uCor Wearers - 1 Year Data
Number analyzed (Participants) | 249 | 96 | 90
score on a scale | 32 (27.1) | 54.8 (28.3) | 58.2 (24.9)

16. Secondary Outcome: Mortality Rate, Heart Failure Related Events, Quality of Life (QoL) and Healthcare Utilization Data at 6 Months and One Year Post Enrollment: Healthcare Utilization Data
Description: For each weekly phone call, monthly office visit, 6-month phone call, and 1-year phone call, each subject reported whether they experienced a hospitalization, emergency room visit, or unplanned doctor's office visit since their last call/visit.
Time Frame: 6 months and 1 year
Population: All subjects in the study from the timepoint of enrollment until end of study participation.
Measure: Number; unit: participants
Groups:
- uCor Wearers - 6 Month Data: All subjects from enrollment until up to 6 months
- uCor Wearers - 1 Year Data: All subjects from enrollment until up to 1 year
Arm/Group | uCor Wearers - 6 Month Data | uCor Wearers - 1 Year Data
Number analyzed (Participants) | 249 | 249
participants
  Subjects with hospitalization for any reason | 120 | 134
  Subjects with ER visit for any reason | 101 | 119
  Subjects with unplanned doctor's office visit for any reason | 55 | 62

ADVERSE EVENTS:
Time Frame: 1 year + 30 days, per subject
Description: All device related adverse effects will be recorded during the study. All adverse device effects (ADEs) will be classified by the investigator as anticipated or unanticipated. Adverse events will also include any adverse events related to medication changes and medical procedures initiated by μCor data.
Groups:
- Single-Arm, Eligible Subjects: Subjects hospitalized for acute decompensated heart failure and enrolled in the study within 10 days post-hospital discharge.
  All subjects require an additional heart failure event within the previous 180 days.
Arm/Group | Single-Arm, Eligible Subjects
All-Cause Mortality (participants affected / at risk) | 37/265
Serious Adverse Events (participants affected / at risk) | 0/265
Other Adverse Events (participants affected / at risk) | 106/265
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Eligible Subjects (N=265)
Skin Irritation (Skin and subcutaneous tissue disorders) | 106 (143)

LIMITATIONS AND CAVEATS:
This study was conducted from 11/1/2019 to 6/30/2023 and partially overlapped with the COVID-19 Pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT04096040/Prot_SAP_000.pdf